CLINICAL TRIAL: NCT03436108
Title: Role of Bisphenol A (BPA) in the Pathogenesis of the Polycystic Ovary Syndrome
Brief Title: Bisphenol Role in the Pathogenesis of PCOS
Status: Completed | Type: Observational
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other); Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Assistant Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: Bisphenol and PCOS
Record Dates: First submitted 2018-02-11; First posted 2018-02-19 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: PCOS
MeSH Terms: interventions — Urination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS group: patients who have PCOS
  Interventions: Diagnostic Test: Measurement of Bisphenol in urine
- control group: patients who donnot have PCOS
  Interventions: Diagnostic Test: Measurement of Bisphenol in urine

INTERVENTIONS:
Diagnostic Test: Measurement of Bisphenol in urine — to see level of this material in blood of women

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common and the most heterogeneous endocrine disorder in premenopausal women. Its prevalence is estimated from 5 to 10% depending on the diagnosis' criteria .

Apart from signs of hyperandrogenism such as acne, hirsutism and hair loss; women with PCOS usually present with menstrual irregularities and fertility problems ..

DETAILED DESCRIPTION:
Bisphenol A is formed from acetone and phenol, it is used in production of epoxy resin, polyster resins and polyvarbonate resins. Epoxy resins are used in plastics, adhesives, and structural composites .

Humans are at the end of the food chain, thus they are exposed to the highest doses of these compounds. EDs have been detected in human adipose tissue and biological fluids such as: serum, urine, milk and amniotic fluid .

Additionally, it has been proven that BPA can also directly stimulate androgen synthesis in the ovarian theca-interstitial cells. A correlation between increased serum testosterone levels observed in women with PCOS with serum BPA concentrations has also been found .

ELIGIBILITY:
Inclusion Criteria:

* Age group: 18-40
* Females
* Diagnosed a case of polycystic ovary syndrome

Exclusion Criteria:

* • Female patients with other acute or chronic illness

  * Cardiovascular disease
  * Neoplasms
  * Current smoking, diabetes mellitus,
  * Renal impairment (serum creatinine 120 mol/liter), and hypertension (blood pressure 140/85 mm Hg).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females with PCOS
Study Population: females who were diagnosed to have PCOS
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
the number of participants who will have high level of bisphenol in btheir blood | within 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt )
Locations (1):
- Algazeerah, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
Results will be shared after finishing the research